CLINICAL TRIAL: NCT07313007
Title: Evaluation of the Production of Amino Acid-Derived Metabolites by the Gut Microbiota of Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Brief Title: Assessment of Gut Microbiota-Derived Amino Acid Metabolite Production in Patients With MASLD
Acronym: MASLD-GUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL25_1015
Record Dates: First submitted 2025-12-11; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolic Dysfunction-Associated Steatohepatitis (MASH)
Keywords: MASLD; MASH; GUT MICROBIOTA; N-acétyl-phenylalanine (NAPA)
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Single-center, non-randomized, prospective, open-label study, with a descriptive and exploratory purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MASLD Group (Other): Patients with metabolic dysfunction-associated steatotic liver disease Participants in this group are adults (18-80 years) with confirmed MASLD based on recent imaging and at least one associated cardiometabolic risk factor. These patients are already monitored in the Endocrinology, Diabetes, and Nutrition Department at Lyon Sud Hospital.
  Interventions: Procedure: stool sampling, dietary assessment, and collection of blood and urine samples
- Healthy Volunteers Group (Other): Healthy volunteers meet the general inclusion criteria shared with the patient group but do not present MASLD or other cardiometabolic diseases and do not have any liver pathology.
  Their participation serves as a control group for comparison with MASLD patients in the context of the study's biological and metabolic analyses.
  Interventions: Procedure: stool sampling, dietary assessment, and collection of blood and urine samples

INTERVENTIONS:
Procedure: stool sampling, dietary assessment, and collection of blood and urine samples — MASLD group includes individuals receiving routine clinical care for liver-related conditions. During their scheduled medical visits, participants undergo standard clinical assessments and routine blood tests. Additional research-specific procedures-such as stool sampling, dietary assessment, and collection of blood and urine samples-are carried out without altering routine patient management. A fraction of blood sample is used for NAPA measurement. Stool samples are collected at home and returned directly to the Endocrinology, Diabetes and Nutrition Department within 24 hours after collection.
  Healthy volunteers undergo the same research-specific procedures as patients but exclusively for research purposes, with no routine-care-related assessments.

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) encompasses a spectrum of liver disorders ranging from simple steatosis-a relatively benign and non-progressive condition-to metabolic dysfunction-associated steatohepatitis (MASH), characterized by hepatocellular inflammation. MASLD is now the leading cause of chronic liver disease worldwide, affecting approximately one in three adults, particularly those with obesity or type 2 diabetes.

Recent studies have highlighted a strong interconnection between the gut microbiota, the liver, metabolism, and the immune system, collectively referred to as the gut-liver axis. Alterations in the gut microbiota are observed at all stages of MASLD, and several microbial metabolites-such as trimethylamine, bile acids, short-chain fatty acids, and ethanol-have been implicated in disease progression.

Emerging evidence points to a role for gut-derived metabolites of tryptophan (Trp) and phenylalanine (Phe), including phenylacetic acid (PAA), 3-(4-hydroxyphenyl)-lactate (HPL), and phenyllactate (PL). These compounds have been associated with the severity of MASLD, particularly with hepatic steatosis and fibrosis. Elevated plasma levels of aromatic amino acids (AAAs), such as L-phenylalanine and L-tyrosine, are also correlated with increased hepatic fat content.

A newly identified Phe-derived metabolite, N-acetyl-phenylalanine (NAPA), together with PAA, HPL, and PL, has been shown to correlate with hepatic steatosis. These metabolites can induce steatosis both in vitro and in vivo, acting through the disruption of endoplasmic reticulum-mitochondria interactions. They therefore represent potential new therapeutic targets.

These four metabolites of interest (NAPA, PAA, HPL, PL) can be produced both by gut bacteria and through endogenous human metabolism. Positive correlations between plasma NAPA concentrations and specific bacterial species have been observed, although the responsible taxa remain to be identified.

HYPOTHESIS

We hypothesize that the gut microbiota of MASLD patients produces aromatic amino acid-derived metabolites, contributing to the elevated plasma concentrations observed in these patients

Two complementary strategies will be used : Human Microbiota Culture and Fecal Microbiota Transplantation

ELIGIBILITY:
Inclusion Criteria:

* For patients and healthy volunteers:

  * Age between 18 and 80 years.
  * Non-diabetic participant (fasting blood glucose < 1.26 g/L, or absence of insulin therapy or oral antidiabetic medication).
  * Body mass index (BMI) between 18 and 30 kg/m².
  * For women of childbearing potential, use of at least one recognized effective contraceptive method.
  * Very regular bowel movements every 24 to 48 hours.
  * Participant living within 100 km of the Lyon Sud Hospital Center (CHLS).
  * Participant willing to participate in the study and providing written informed consent.
  * Participant affiliated with the general French Social Security system or an equivalent scheme.
* For patients:

  * Presence of MASLD according to the definition of the European Association for the Study of the Liver (EASL), defined by hepatic steatosis on imaging performed within the previous year (abdominal ultrasound, abdominal CT scan, magnetic resonance imaging, or controlled attenuation parameter (CAP) measured by FibroScan) and at least one cardiometabolic criterion among: dyslipidemia, arterial hypertension, overweight (BMI ≥ 25 kg/m²), impaired glucose tolerance, or type 2 diabetes.
  * No history of liver transplantation.
  * No excessive alcohol consumption (less than 20 g/day for women and less than 30 g/day for men).
  * Patient followed in the Endocrinology, Diabetes and Nutrition Department at Lyon Sud Hospital.

Exclusion Criteria:

* For patients and healthy volunteers:

  * Participant with active inflammatory, infectious, cardiovascular, or neoplastic disease.
  * Participant with a history of colectomy, small bowel resection, or cholecystectomy.
  * Participant who received antibiotics, prebiotics, or probiotics within the past 3 months.
  * Participant using laxatives (more than 2 doses per day over the past 3 months).
  * Participant with chronic constipation.
  * Pregnant, parturient, or breastfeeding women.
  * Participant deprived of liberty by judicial or administrative decision.
  * Participant receiving psychiatric care.
  * Participant institutionalized for reasons other than research.
  * Adult participant under legal protection (guardianship or trusteeship).
  * Participant who does not understand the French language and cannot provide informed consent.
  * Participant already enrolled in a study presenting a conflict of interest with the present study.
* For healthy volunteers

  * Known liver disease
  * No long-term drug medication except oral contraception for women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of NAPA in Stool Culture Medium | Within 30 days after Visit 1 (sample collection and analysis performed at a single time point)
  Quantification of the metabolite N-acetyl-phenylalanine (NAPA) in the culture medium of stool samples cultivated using the MiPro in vitro human gut microbiota culture system.

SECONDARY OUTCOMES:
Concentration of Selected AAA-Derived Metabolites in Stool Culture Medium | Within 30 days after Visit 1 (sample collection and analysis performed at a single time point)
  Quantification of selected aromatic amino acid (AAA)-derived metabolites in the culture medium of stool samples cultivated using the MiPro in vitro human gut microbiota culture system.
Gut Microbiota Composition in Stool Samples | Within 30 days after Visit 1 (sample collection and analysis performed at a single time point)
  Characterization of gut microbiota composition in stool samples who produce NAPA or other metabolites of interest, to identify bacterial species potentially involved in metabolite production. Microbiota profiling will be performed on a stool sample using bacterial DNA sequencing methods (16S rRNA gene sequencing or shotgun metagenomics).
Concentration of NAPA in plasma | Baseline Visit 1 (sample collection and analysis performed at a single time point)
  The quantification of NAPA level will be performed on plasma samples

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud Service Endocrinologie, Diabète et nutrition, Pierre-Bénite, France